CLINICAL TRIAL: NCT06648746
Title: Predictors of Therapeutic Success and Adverse Events in Endoscopic Ampullectomy
Status: Not yet recruiting | Type: Observational
Sponsor: Universidade do Porto (Other)
Responsible Party: Principal Investigator, Paulo Sérgio Durão Salgueiro, MD, PhD, Universidade do Porto
Other Study IDs: 112233
Record Dates: First submitted 2024-10-14; First posted 2024-10-18 (Actual); Last update posted 2024-10-18 (Actual); Status verified 2024-10

CONDITIONS: Ampulla of Vater Adenoma; Ampulla of Vater Disease (Benign/Malignancy)
MeSH Terms: conditions — Neoplasms

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Endoscopic ampullectomy: Consecutive adult patients submitted to endoscopic resection of an ampullary adenoma in each of the participating center for which endoscopic ampullectomy was performed from 1st January 2019 to 31th December will be included. Clinical and demographic data related to the patient, and data pertaining to the ampullary lesion and the endoscopic ampullectomy procedure will be obtained by reviewing the medical records of each participating center.

SUMMARY:
Although ampullary tumors are rare (representing 0.6-0.8 % of all digestive cancers), their estimated incidence has increased in recent years (<1 per 100 000 per year). Most noninvasive ampullary tumors of the major papilla occur as sporadic and asymptomatic lesions, detected during conventional upper endoscopy performed for another indication.

Nonetheless, they can present with jaundice (17%), pain (14%), pancreatitis (4%), cholangitis (1%), and can be associated with common bile duct stones (up to 38%). Resection of ampullary adenomas is warranted to prevent malignant progression. The most recent European Society of Gastrointestinal Endoscopy (ESGE) recommend endoscopic ampullectomy as the standard of care approach for ampullary adenomas without intraductal extension, due to excellent outcomes of technical and clinical success (high complete and curative resection rates of 94% and 87%, respectively), with lower morbidity and recurrence rates. This procedure as a low rate of mortality (of 0.4%), but the rate of adverse events can exceed 20%. The most frequent adverse events are acute pancreatitis (12%), intraprocedural and/or delayed bleeding (11%), perforation (3%), cholangitis (3%), ampullary stenosis (2.5%). Also there is a high recurrence rate of up to one third after endoscopic resection; up to two thirds are identified at the first follow-up endoscopy, requiring additional endoscopic resection or surgery.

DETAILED DESCRIPTION:
The relevance of the study is to assess the predictors for therapeutic success, adverse events and recurrence after endoscopic ampullectomy is of paramount importance to develop expertise in this challenging procedure.

The occurrence of adverse events after endoscopic ampullectomy carries a significant impact on the prognosis and recovery, possibly limiting a broader proficiency in this procedure. Thus, identifying significant predictors is crucial to more accurately select the patients and to evolve strategies to prevent and minimize the incidence and severity of adverse events.

ELIGIBILITY:
Inclusion Criteria:

* Adult patients (≥18 years) submitted to endoscopic resection of an ampullary adenoma with the following features were included:

  * lesions up to 30 mm (including with laterally spreading component)
  * with low-grade or high-grade dysplasia on preprocedural histology
  * with no intraductal extension
  * with no evidence of invasive malignancy on endoscopic assessment (including endoscopic features including hard consistency, friable or ulcera:ve surface and spontaneous bleeding)
* A minimum follow-up period of one year afer endoscopic ampullary resection.

Exclusion Criteria:

* Patients with lesions with the following features were excluded:

  * intraductal extension
  * evidence of invasive malignancy
  * other non-adenomatous lesions
* Patients who underwent endoscopic resection or surgical ampullectomy prior to enrollment
* Patients with a follow-up of less than a year after endoscopic ampullary resection
* Patients with pancreas divisum.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Consecutive adult patients submihed to endoscopic resection of an ampullary adenoma in each of the participating center (ULS de Santo António - Porto; ULS São João - Porto)
Sampling Method: Non-Probability Sample
Enrollment: 100 (Estimated)
Dates: Start 2024-12 (Estimated); Primary Completion 2024-12 (Estimated); Study Completion 2024-12 (Estimated)

PRIMARY OUTCOMES:
Therapeutic success | 1 year
  - Rate of adenoma recurrence after endoscopic resection of ampullary adenomas
Safety outcomes | 1 year
  - Rate of adverse events related to endoscopic resection of ampullary adenomas

SECONDARY OUTCOMES:
Prophylaxis | 1 year
  - Comparison of the post-ampullectomy acute pancreatitis incidence with different kinds of prophylaxis
Risk factors | 1 year
  To perform a multivariate analysis of patient, lesion and procedure characteristics that correlate with the incidence of adverse events

CONTACTS AND LOCATIONS:
Overall Officials: Paulo Salgueiro, MD, PhD, Principal Investigator — Universidade do Porto

IPD SHARING:
Plan to Share IPD: Undecided
Not decided yet

REFERENCES:
- [Background] Walter D, Schnitzbauer AA, Schulze F, Trojan J. The Diagnosis and Treatment of Ampullary Carcinoma. Dtsch Arztebl Int. 2023 Oct 27;120(43):729-735. doi: 10.3238/arztebl.m2023.0195. PMID 37656482
- [Background] Vanbiervliet G, Strijker M, Arvanitakis M, Aelvoet A, Arnelo U, Beyna T, Busch O, Deprez PH, Kunovsky L, Larghi A, Manes G, Moss A, Napoleon B, Nayar M, Perez-Cuadrado-Robles E, Seewald S, Barthet M, van Hooft JE. Endoscopic management of ampullary tumors: European Society of Gastrointestinal Endoscopy (ESGE) Guideline. Endoscopy. 2021 Apr;53(4):429-448. doi: 10.1055/a-1397-3198. Epub 2021 Mar 16. PMID 33728632
- [Background] Shahzad MI, Pickering G, Zafar M, Hayat S, Vlavianos P. The Duodenal Accessory Ampulloma and the Role of Endoscopic Retrograde Cholangiopancreatography (ERCP) in Familial Adenomatous Polyposis Coli Inheritance. Cureus. 2024 May 1;16(5):e59445. doi: 10.7759/cureus.59445. eCollection 2024 May. PMID 38826909
- [Background] Rizzo A, Dadduzio V, Lombardi L, Ricci AD, Gadaleta-Caldarola G. Ampullary Carcinoma: An Overview of a Rare Entity and Discussion of Current and Future Therapeutic Challenges. Curr Oncol. 2021 Sep 1;28(5):3393-3402. doi: 10.3390/curroncol28050293. PMID 34590592
- [Background] Poley JW, Campos S. Methods and outcome of the endoscopic treatment of ampullary tumors. Ther Adv Gastrointest Endosc. 2020 Jan 21;13:2631774519899786. doi: 10.1177/2631774519899786. eCollection 2020 Jan-Dec. PMID 32030370
- [Background] Patel R, Varadarajulu S, Wilcox CM. Endoscopic ampullectomy: techniques and outcomes. J Clin Gastroenterol. 2012 Jan;46(1):8-15. doi: 10.1097/MCG.0b013e318233a844. PMID 22064552
- [Background] Maselli R, de Sire R, Fugazza A, Spadaccini M, Colombo M, Capogreco A, Beyna T, Repici A. Updates on the Management of Ampullary Neoplastic Lesions. Diagnostics (Basel). 2023 Oct 6;13(19):3138. doi: 10.3390/diagnostics13193138. PMID 37835881
- [Background] Lai JH, Shyr YM, Wang SE. Ampullectomy versus pancreaticoduodenectomy for ampullary tumors. J Chin Med Assoc. 2015 Jun;78(6):339-44. doi: 10.1016/j.jcma.2015.02.002. Epub 2015 Mar 26. PMID 25818543
- [Background] Klair JS, Irani S, Kozarek R. Best techniques for endoscopic ampullectomy. Curr Opin Gastroenterol. 2020 Sep;36(5):385-392. doi: 10.1097/MOG.0000000000000657. PMID 32740000
- [Background] Kim AL, Choi YI. Safety of duodenal ampullectomy for benign periampullary tumors. Ann Hepatobiliary Pancreat Surg. 2017 Aug;21(3):146-150. doi: 10.14701/ahbps.2017.21.3.146. Epub 2017 Aug 31. PMID 28990001
- [Background] Jung YK, Paik SS, Choi D, Lee KG. Transduodenal ampullectomy for ampullary tumor. Asian J Surg. 2021 May;44(5):723-729. doi: 10.1016/j.asjsur.2020.12.021. Epub 2021 Jan 21. PMID 33485767
- [Background] Jiang L, Chai N, Li M, Linghu E. Therapeutic Outcomes and Risk Factors for Complications of Endoscopic Papillectomy: A Retrospective Analysis of a Single-Center Study. Ther Clin Risk Manag. 2021 May 28;17:531-541. doi: 10.2147/TCRM.S309103. eCollection 2021. PMID 34093018
- [Background] Dumonceau JM, Kapral C, Aabakken L, Papanikolaou IS, Tringali A, Vanbiervliet G, Beyna T, Dinis-Ribeiro M, Hritz I, Mariani A, Paspatis G, Radaelli F, Lakhtakia S, Veitch AM, van Hooft JE. ERCP-related adverse events: European Society of Gastrointestinal Endoscopy (ESGE) Guideline. Endoscopy. 2020 Feb;52(2):127-149. doi: 10.1055/a-1075-4080. Epub 2019 Dec 20. PMID 31863440
- [Background] Choi SJ, Lee HS, Kim J, Choe JW, Lee JM, Hyun JJ, Yoon JH, Kim HJ, Kim JS, Choi HS. Clinical outcomes of endoscopic papillectomy of ampullary adenoma: A multi-center study. World J Gastroenterol. 2022 May 7;28(17):1845-1859. doi: 10.3748/wjg.v28.i17.1845. PMID 35633905
- [Background] Alali A, Espino A, Moris M, Martel M, Schwartz I, Cirocco M, Streutker C, Mosko J, Kortan P, Barkun A, May GR. Endoscopic Resection of Ampullary Tumours: Long-term Outcomes and Adverse Events. J Can Assoc Gastroenterol. 2020 Feb;3(1):17-25. doi: 10.1093/jcag/gwz007. Epub 2019 Mar 18. PMID 32010876